CLINICAL TRIAL: NCT01964677
Title: Magnetic Resonance-Guided High Intensity Focused Ultrasound for Palliation of Painful Skeletal Metastases - a Multicenter Study
Brief Title: MR-HIFU for Bone Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Principal Investigator, NdeSouza, Professor of Translational Imaging, Institute of Cancer Research, United Kingdom
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12/LO/0424 CCR3772
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cancer; Bone Metastases
Keywords: Magnetic Resonance Imaging (MRI); High Intensity Focused Ultrasound (HIFU)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MR-HIFU of painful bone metastases (Experimental)
  Interventions: Device: Magnetic Resonance Image-guided High Intensity Focused Ultrasound (MR-HIFU)

INTERVENTIONS:
Device: Magnetic Resonance Image-guided High Intensity Focused Ultrasound (MR-HIFU)

SUMMARY:
The aim of this study is to evaluate effectiveness of the Philips Sonalleve MR-HIFU device for the palliation of pain in patients with bone metastases.

Magnetic Resonance Imaging-guided High Intensity Focused Ultrasound (MR-HIFU) uses ultrasound to palliate pain caused by bone metastases. The main palliative mechanism of the method is due to local bone denervation, caused by the heat denaturation of the periosteum layer in the treated area. The importance of this therapy is that it offers a non-invasive, focal therapy, avoiding side-effects to surrounding normal tissue that occur with radiation therapy or the need for needle insertion as with radio-frequency(RF)ablation.

The study hypothesis is that MR-HIFU will be effective in treating the pain associated with bone metastases

ELIGIBILITY:
Inclusion Criteria:

* radiologic evidence of bone metastases from any solid tumour
* diagnosis of dominant painful bone metastasis
* target lesion less than 8cm

Exclusion Criteria:

* primary bone tumours rather than metastases
* Inability to tolerate stationary position during treatment
* pregnancy
* MRI incompatible metal implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Pain response | 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nandita deSouza, Professor, Principal Investigator — ICR
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom